CLINICAL TRIAL: NCT06123884
Title: A Phase II/III Study to Evaluate the Safety and Efficacy of BAT1308 Combined with Platinum-Based Chemotherapy ± Bevacizumab As First-Line Therapy for PD-L1-Positive (CPS ≥ 1) Persistent, Recurrent or Metastatic Cervical Cancer
Brief Title: BAT1308 Combined with Platinum-Based Chemotherapy± Bevacizumab for PDL1-Positive (CPS ≥1) Cervical Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BAT-1308-002-CR
Record Dates: First submitted 2023-09-21; First posted 2023-11-09 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Bevacizumab; Carboplatin; Paclitaxel; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BAT1308 (Experimental): Strength 100 mg/4 mL, intravenous drip, recommended dose 300 mg, administered every 3 weeks (21 days) (Q3W)
  Interventions: Drug: Recombinant humanized anti-PD-1 monoclonal antibody injection; Drug: Cisplatin; Drug: Bevacizumab Injection; Drug: carboplatin; Drug: Paclitaxel for Injection
- BAT1308 monoclonal antibody (Placebo Comparator): Strength 100 mg/4 mL, intravenous drip, recommended dose 300 mg, administered every 3 weeks (21 days) (Q3W)
  Interventions: Drug: Recombinant humanized anti-PD-1 monoclonal antibody injection; Drug: Cisplatin; Drug: Bevacizumab Injection; Drug: carboplatin; Drug: Paclitaxel for Injection

INTERVENTIONS:
Drug: Recombinant humanized anti-PD-1 monoclonal antibody injection — Strength 100 mg/4 mL, intravenous drip, recommended dose 300 mg, administered every 3 weeks (21 days) (Q3W).
  Other Names: BAT1308 injection
Drug: Cisplatin — the usage and dosage should be determined by the investigator
  Other Names: Shunbo
Drug: Bevacizumab Injection — Strength 100 mg/4 mL, recommended dose 15 mg/kg body weight, administered every 3 weeks (15 mg/kg, Q3W)
  Other Names: Pobevcy
Drug: carboplatin — the usage and dosage should be determined by the investigator
  Other Names: Bobei
Drug: Paclitaxel for Injection — the usage and dosage should be determined by the investigator
  Other Names: Tesu

SUMMARY:
Phase II study: a study to explore the safety and preliminary efficacy of BAT1308 combined with platinum-based chemotherapy ± Bevacizumab Phase III study: a confirmatory study to evaluate the safety and efficacy of BAT1308 combined with platinum-based chemotherapy ± Bevacizumab as first-line therapy for PD-L1-positive (CPS ≥ 1) persistent, recurrent or metastatic cervical cancer

DETAILED DESCRIPTION:
The single-arm Phase II exploratory study designed to evaluate the safety and efficacy of the study drug will include 20-50 subjects to explore the safety and preliminary efficacy of BAT1308 combined with platinum-based chemotherapy ± Bevacizumab. Dynamic analysis will be conducted after the inclusion of 20 subject. If the safety of this combination regimen is manageable and the efficacy meets expectations, the enrollment in the Phase II study will be stopped and the Phase III study will be entered. The Phase III study is a randomized, double-blind, multicenter clinical study of BAT1308 combined with platinum-based chemotherapy ± Bevacizumab versus placebo plus platinum-based chemotherapy ± Bevacizumab as first-line therapy for PD-L1-positive (CPS ≥ 1) persistent, recurrent or metastatic cervical cancer. PFS and OS will be used as the combined endpoints, and a superiority design will be adopted with a total sample size of 476 subjects. Stratified block randomization will be performed based on the following random factors: patients will be stratified based on the presence of metastatic diseases at the time of diagnosis (Yes vs. No), PD-L1 CPS (1-10 vs. ≥ 10) and planned use of Bevacizumab (Yes vs. No).

ELIGIBILITY:
inclusion criteria：

1. Female patients, aged ≥18 years to ≤70 years, who voluntarily sign the informed consent form;
2. With persistent, recurrent or metastatic (the Federation International of Gynecology and Obstetrics [FIGO] Stage IVB) cervical cancer confirmed histologically (pathological reports required), including pathological types of squamous cell carcinoma, adenocarcinoma, adenosquamous cell carcinoma and clear-cell renal-cell carcinoma, not amenable to radical surgery and/or radical radiotherapy or radiochemotherapy, with no prior systemic anti-tumor therapy for persistent, recurrent or metastatic cervical cancer;
3. Subjects should be positive for PD-L1 expression (CPS ≥ 1) in tumor specimens by the central laboratory. Subjects should provide sufficient formalin-fixed paraffin-embedded (FFPE) specimens or sections (6 sections recommended, not less than 3 sections), and be willing to undergo a tumor tissue biopsy for PD-L1 testing when necessary. The archival tissues must be representative tumor specimens collected within three years or unstained continuous sections of FFPE tumor tissues freshly resected within six months, and relevant pathological reports of the aforementioned specimens must also be provided. Both surgical resection and biopsy are acceptable methods for acquiring fresh tissue specimens; fine-needle aspiration and liquid-based cytology (TCT) samples (i.e., samples lacking complete tissue structures and providing only cell suspension and/or cell smears) are not acceptable; decalcified bone metastasis tumor tissue specimens are not acceptable;
4. At least one measurable tumor lesion per RECIST v1.1; lesions at sites previously treated with radiotherapy or other loco-regional therapies can only be considered as non-target lesions, unless unequivocal progression of the lesion occurs or the tumor activity of the lesion is confirmed by biopsy and the lesion is measurable
5. Life expectancy ≥12 weeks as evaluated by the investigator;
6. Eastern Cooperative Oncology Group (ECOG) Performance Status score 0 or 1;
7. Female patients of childbearing potential must have a negative serum pregnancy test within 7 days before the first dose and are willing to take effective birth control/contraceptive methods to prevent pregnancy during the study until 6 months after the last dose of the study drug. Postmenopausal women must have amenorrhea for at least 12 months before they are considered as women of non-childbearing potential.

9. Able to understand trial requirements, willing and able to comply with the trial and follow-up procedures.

exclusion criteria：

1. Subjects with other pathological types of cervical cancer, such as small cell carcinoma, sarcoma, etc.;
2. Pregnant or lactating women;
3. Prior radiotherapy within 14 days before the first dose. Except for palliative area radiotherapy for bone metastases for which pain cannot be effectively controlled by systemic therapy or local pain relief (radiotherapy area < 5% of bone marrow area); prior chemotherapeutic agents for increasing the sensitization to radiotherapy within 14 days before the first dose; prior use of traditional Chinese patent medicines or treatment with anti-tumor related functions as specified in the NMPA-approved package inserts within 14 days before the first dose, or Chinese herbal medicines for anti-tumor purposes clearly documented in the medical record ;
4. Patients who received live/attenuated vaccines and mRNA vaccines within 4 weeks prior to screening or scheduled to receive those vaccines during the study period;
5. Any prior treatments targeting the mechanism of tumor immunity, such as immune checkpoint inhibitors (e.g., anti-PD-1 antibodies, anti-PD-L1 antibodies, anti-CTLA-4 antibodies, etc.) or therapies that target immune co-stimulatory molecules (e.g., antibodies targeting ICOS, CD40, CD137, GITR, OX40, etc.);
6. AEs caused by prior anti-tumor therapy that are still > Grade 1 (as per CTCAE v5.0) before the first dose of the study drug (except for AEs, such as alopecia, fatigue, etc., that cannot be recovered to ≤ Grade 1 and will remain stable for a long time as judged by the investigator based on actual clinical situations, except for Grade 2 peripheral neurotoxicity, and hypothyroidism stabilized by hormone replacement therapy); patients who previously experienced ≥ Grade 3 irAEs or discontinued immunotherapy due to irAEs of any grade;
7. Active leptomeningeal disease or poorly controlled brain metastases. Patients with suspected or confirmed brain metastases are allowed to be enrolled if they have no obvious symptoms and the results of imaging examinations performed at least 28 days before the first dose of the study drug showed stable disease and no treatment (e.g., radiotherapy, surgery, or corticosteroid treatment) is required to control the symptoms of brain metastases within 28 days before the first dose of the study drug;
8. Patients who underwent major organ surgery (excluding aspiration biopsy) or experienced significant trauma within 4 weeks before the first dose of the study drug, or those who require elective surgery during the trial period;
9. Subjects with serious infections within 4 weeks before the first dose, including but not limited to the infection-related complications, bacteremia and severe pneumonia requiring hospitalization; subjects with active infection before the first dose are excluded;
10. Patients with the following infectious diseases: human immunodeficiency virus (HIV) infection; active hepatitis B virus infection [hepatitis B surface antigen (HBsAg) positive, and the result for hepatitis B virus deoxyribonucleic acid (HBV-DNA) test > 500 IU/ml or 103 copies/ml or above the upper limit of normal at the testing institution]; hepatitis C virus infection [anti-HCV antibodies and hepatitis C virus ribonucleic acid (HCV-RNA) test positive]; Treponema pallidum antibody positive and rapid plasma reagin (RPR) positive;
11. Subjects with tuberculosis untreated or under treatment, including but not limited to pulmonary tuberculosis; patients whose tuberculosis was cured after standardized anti-tuberculosis treatment as confirmed by the investigator may be included;
12. Subjects with known history of severe allergy or prior ≥ Grade 3 allergic reactions to macromolecular protein preparations/monoclonal antibodies, and any component of the investigational drug;
13. Known to have any contraindication to cisplatin/carboplatin or paclitaxel, or allergy to any of their components;
14. Clinically significant hydronephrosis that cannot be relieved by nephrostomy or ureteral stent insertion as judged by the investigator;
15. Subjects with uncontrollable pleural effusion, pericardial effusion, or ascites requiring repeated drainage;
16. Patients with active or potentially recurrent autoimmune disease (excluding patients with vitiligo, autoimmune thyroid disorder that can be treated with hormone replacement therapy, or type 1 diabetes mellitus);
17. Patients who required systemic treatment with glucocorticoid (>10 mg/day of prednisone or equivalent) or other immunosuppressive agents within 14 days before the first dose of the study drug, except for the following situations: ① topical, ocular, intra-articular, nasal, and inhaled glucocorticoid therapy; ② short-term use of glucocorticoid for prophylaxis (e.g., prevention of contrast allergy);
18. Subjects with a history of noninfectious pneumonitis requiring glucocorticoid therapy within 1 year before the first dose or with current interstitial lung disease;
19. History of severe cardiovascular and cerebrovascular disorders, including but not limited to: ① New York Heart Association (NYHA) Class II or above cardiac failure or left ventricular ejection fraction (LVEF) <50%; ② Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, II-III degree atrioventricular block, etc.; ③ Acute coronary syndrome, congestive cardiac failure, aortic dissection, stroke, or other Grade 3 or above cardiovascular and cerebrovascular events within 6 months before the first dose; ④ Clinically uncontrollable hypertension (defined in this protocol as systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg despite the use of antihypertensive therapy);

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From first administration to the occurrence of objective tumor progression or all-cause death (whichever occurs first), the assessment period lasts up to two years.
  Tumor assessment is performed according to RECIST 1.1. Tumor imaging assessment is performed every 9 weeks (±7 days) after the first administration until week 54. After that, it is performed once every 12 weeks (±7 days) until disease progression, withdrawal from the group, loss to follow-up, death, or 24 months after the first study drug administration at the longest distance, whichever occurs first.
Overall Survival | From the date of first administration to the time of death due to any cause, the assessment period will last up to two years.
  Tumor assessment is performed according to RECIST 1.1. Tumor imaging assessment is performed every 9 weeks (±7 days) after the first administration until week 54. After that, it is performed once every 12 weeks (±7 days) until disease progression, withdrawal from the group, loss to follow-up, death, or 24 months after the first study drug administration at the longest distance, whichever occurs first.

SECONDARY OUTCOMES:
Vital signs | Through study completion, an average of 2 years
  Number of cases with abnormal vital signs results
Physical examination | Through study completion, an average of 2 years
  Number of cases with abnormal physical examination results
Laboratory Examination | Through study completion, an average of 2 years
  Number of cases with abnormal laboratory examination results
Adverse event | Through study completion, an average of 2 years
  Number of cases with all adverse medical events that occur after the subject receives the investigational drug assessed by CTCAE V5.0
Objective response rate (ORR) | Through study completion, an average of 2 years
  The proportion of subjects whose tumors have shrunk by a certain amount and remained so for a certain period of time.
anti-drug antibodies | cycle1,cycle3,cycle5 and every 9 weeks after cycle5, 21 days is a cycle and the evaluation lasts for up to 2 years.
  All subjects need to collect blood samples at specific time points during the treatment period. At each time point, about 4.0 mL of blood sample is planned to be collected to detect anti-drug antibodies
neutralizing antibody | cycle1,cycle3,cycle5 and every 9 weeks after cycle5, 21 days is a cycle and the evaluation lasts for up to 2 years.
  All subjects need to collect blood samples at specific time points during the treatment period. At each time point, about 4.0 mL of blood sample is planned to be collected to detect neutralizing antibody

CONTACTS AND LOCATIONS:
Overall Officials: Qinglei Gao, Ph.D, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei, China